CLINICAL TRIAL: NCT01771159
Title: Tissue Bonding Cystostomy(TBC)
Acronym: TBC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uro-Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Spinal Cord Injury (SCI); Chronic Urinary Retention; Urinary Incontinence
Keywords: Spinal cord injury; Urinary dysfunction; Bladder drainage
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Population (Experimental): All subjects will undergo the implantation of the TBC.
  Interventions: Device: TBC

INTERVENTIONS:
Device: TBC — The anchor is capped and surgically implanted in the extra-peritoneal space of the suprapubic region of pubic hair of the lower abdomen using sutures sandwich and secure the anchor between the rectus abdominis muscle and the detrusor [bladder] muscle. Skin is closed over the implant and the bladder is drained with a Foley urethral catheter. The Phase I implant is left in place for 3+ months to allow fibroblasts and collagen from the adjacent muscles to grow into the porous PTFE and effect robust, water--tight bonding of anchor to both rectus and bladder muscles.
  After a local anesthesia is injected, the remaining components of the TBC are connected forming a water-tight union of the anchor to the urinary bladder.

SUMMARY:
Spinal Cord Injured [SCI] patients typically cannot "pee". Injury to the spinal cord disrupts the in-coming and out-going brain signals that coordinate bladder sensation and the emptying of bladder. SCI typically causes chronic retention of urine with uncontrolled leakage of urine. Some form of tube (catheter) is needed to drain the urine except with the mildest forms of SCI. Two types of tubes to drain the urine have been used for many years. These types are the urethral (inserted into the bladder through the opening usually used to empty the bladder) and abdominal, called suprapubic cystostomy tubes (put into the bladder through the abdomen).

Bacteria (germs) normally live on our skin. Bacteria have sticky surfaces and so they stick to catheter surfaces. Bacteria reproduce very rapidly from a few dozen to over a million in 24 hours. In a warm liquid environment, like urine, bacteria can reach a density of 10 million per cubic centimeter in 48 hours which causes infection. Oral drugs and antibiotic-coated catheters delay this process by a week or two, but within a month 100% of patients have bacteria in their urine. Existing drugs cannot eliminate these microbial sanctuaries.

The TBC is a 'closed access' abdominal drainage tube that has a 'cuff' or 'anchor'. It is permanently placed in the abdominal muscle to bond with the body's tissue. Another catheter is temporarily connected to the TBC that is easily replaceable in the clinic without anesthesia or special instruments. It locks to form a water-tight system. Many parts of the TBC are coated with an antibacterial substance that will delay the growth of bacteria. The TBC has been used with success in multiple animal studies.

This is a Phase I human clinical trial in which the TBC will be used 10 spinal cord injured patients, each of whom will be followed for 12 months or longer. Abdominal catheter exit sites will be photographed monthly and tested periodically to document growth of any bacteria. Every three months, patients will complete satisfaction questionnaires and their urine will be tested for bacteria. Urine will also be tested as clinically indicated.

DETAILED DESCRIPTION:
Traumatic spinal cord injury (SCI) results in permanent paraplegia or quadriplegia in approximately 10,000 Americans annually. All patients with SCI have neuropathic dysfunction of the urinary bladder. Progressive neurological syndromes such as multiple sclerosis, Parkinson's disease, Stroke, hemiplegia and dementia also induce progressive neuropathic bladder dysfunction. Neurologic impairment of the bladder causes or contributes to chronic urinary retention or urinary incontinence or both. Several million Americans suffer chronic neuropathic urinary retention or incontinence or both. Males tend to develop urinary retention and females tend to develop urinary incontinence but both genders commonly develop elements of both.

Current management includes [a] indwelling tubes (urethral catheterization or [b] suprapubic (abdominal) catheterization, [c] intermittent urethral catheterization [4+times per day], and surgical rehabilitation [e.g. use of autogenous intestinal conduits or reservoirs]. No single form of management is ideal. A high percentage of elder and disabled patients are poor candidates or non-candidates for surgical rehabilitation because of co-morbidities or limited life expectancy. A majority of neurologically impaired patients are managed with chronic tube drainage of their bladders [e.g. a-c, above].

Traditional tube drainage of the bladder may be either via the urethra or via an intubated fistula in the lower abdomen. Intermittent catheterization-by the patient or a care giver--via the urethra is a well accepted and sometimes used method. This technique is occasionally used [by an attendant] in cognitively impaired patients or quadriplegics with impairment of the upper extremities. Intermittent catheterization is expensive when provided by a professional care giver and is a social and domestic burden when provided by a family member. In most chronically impaired [cognitively or physically] patients chronic indwelling urethral or suprapubic tubes evolve as the most practical and widely used treatment option.

Chronic urinary infection and bladder stones are recurrent problems in patients who use indwelling tubes. Foley urethral catheters [which are also commonly used as suprapubic tubes] are licensed for 30 day use by FDA.

Indwelling urethral catheters and suprapubic tubes are "open eco-systems' and provide easy access to skin flora. Skin microbes migrate along the tubes and gain access to bladder urine which becomes colonized in 100% of cases. Both gram-stain positive [gram +] and gram-stain negative [gram-] organisms easily gain access to bladder urine. Both type of microbes form biofilms on the catheters within 48 hours of colonization. The biofilms are microbial sanctuaries that are highly resistant to eradication with antibiotics. Use of antimicrobial agents [often for non-urinary indications] may eradicate common urinary pathogens and thereby 'select' more resistant organisms. Multiple organisms and resistant organisms are commonly grown from the bladders of neurologically impaired patients who utilize indwelling urethral or suprapubic tubes. Both types of tubes tend to induce bladder spasms and urinary leakage thereby soiling under-garments and bed clothes. A majority of such patients smell of urine-chronically.

Urine is normally supersaturated with dissolved salts, notably physiologic concentrations of calcium, phosphorus, oxalic acid, and magnesium. Foreign bodies [e.g. the indwelling tube'] initiate nucleation of the salts which then precipitate and form stones on the catheters. A high percentage of neurologically impaired patients have Proteus species of chronic bacteriuria. These urea-splitting [urease producing] organisms greatly accelerate formation of struvite [magnesium-ammonium-phosphate] stones on the catheters; rapid stone formation may necessitate catheter exchanges more frequently than monthly.

Significant expense attends the chronic use of traditional urinary catheters. Monthly travel to clinics and monthly replacement of the drainage catheter and management of febrile reactions which may be precipitated by tube changes are routine and expensive. Surgical procedures are commonly required to remove bladder, kidney or ureteral stones that develop as a consequence of the chronic bacteriuria. Soiled garments and beds and the prevailing order of urine cause many disabled patients to be put in to assisted care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older that have spinal cord injury and/or chronic, irreversible neuropathic bladder dysfunction from other progressive neurological syndromes including Stroke, multiple sclerosis and Parkinsonism.
* Candidates must have a minimum duration of injury and bladder dysfunction of 2 years
* Candidates shall be those who utilize:

  * an indwelling Foley catheter,
  * an indwelling suprapubic catheter,
  * diapers or
  * external (condom) catheter drainage or intermittent self-catheterization but finds the current alternative to be socially unsatisfactory.
* Candidates need to recognize the investigational nature of the "tissue bonding cystostomy" device and must be willing to return for periodic follow-up.
* Candidates also need to recognize that a minor surgical procedure may be needed to remove the device if it proves unsatisfactory.
* Patients must be willing and capable of signing the Informed Consent Document (ICD).
* In the feasibility study detailed in this protocol only English-speaking subjects will be accepted for participation. If the protocol is expanded then a Spanish-language consent form will be developed and Spanish-speaking candidates will be accepted.

Exclusion Criteria:

* have a reversible spinal cord injury or a reversible neurological illness
* have been injured less than two years
* have acceptable forms of urological management utilizing intermittent self-catheterization, or
* spontaneous voiding with the use of an external collecting appliance.
* have no advanced neuropathic bladder dysfunction of less than 2 years duration
* have advanced neuropathic bladder dysfunction and are happy with intermittent self-catheterization or more traditional forms of tube drainage are non-candidates.
* This feasibility study will exclude females of child-bearing age. In subsequent expanded clinical trials it may be appropriate [depending on the outcome of the feasibility study] to include females of child-bearing age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-05; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Continuous use | 12 months
  Continuous use and function of the anchor component for 1+ years following activation

SECONDARY OUTCOMES:
Chronic microbial colonization | 12 months
  Secondary success is defined as elimination of chronic microbial colonization of urine on three of four follow-up urine cultures made during the planned 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P. Smith, MD, Principal Investigator — Baylor College of Medicine